CLINICAL TRIAL: NCT05862233
Title: A Phase Ⅲ Clinical Study to Evaluate the Safety and Efficacy of MIL62 Injection in Participants With Primary Membranous Nephropathy
Brief Title: A Phase Ⅲ Clinical Study of MIL62 in Primary Membranous Nephropathy
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Beijing Mabworks Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIL62-CT307
Record Dates: First submitted 2023-05-08; First posted 2023-05-17 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-10

CONDITIONS: Primary Membranous Nephropathy
MeSH Terms: interventions — Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIL62 (Experimental)
  Interventions: Drug: MIL62
- Cyclosporine (Active Comparator)
  Interventions: Drug: Cyclosporine

INTERVENTIONS:
Drug: MIL62 — An intravenous (IV) infusion of 1000 mg of MIL62 will be administered at Week 1 and Week 3.If the treatment is effective, MIL62 will continue be administered at W25 and W27
  Arms: MIL62
Drug: Cyclosporine — Participants will receive Cyclosporine at a starting oral dose 3.5 mg/kg/d in 2 divided doses, try to give every 12 hours.The dose was adjusted according to the blood concentration of cyclosporine monitored every 2 weeks±3 days until the target blood concentration of 125~175 ng/mL was reached.Optimized cyclosporine dose will be maintained for a maximum 52 weeks dependent on response and then tapered over 8 weeks.
  Arms: Cyclosporine

SUMMARY:
This study will evaluate the efficacy, safety, pharmacokinetics(PK) ,pharmacodynamics（PD）and anti-drug antibodies（ADA） of MIL62 compared with cyclosporine in participants with primary membranous nephropathy (pMN).

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-80;
2. Diagnosis of primary membranous nephropathy (pMN) according to renal biopsy prior to or during screening;
3. Screening 24-hour urinary protein >= 5 g after best supportive care for >= 3 months prior to screening or screening Screening 24-hour urinary protein > 3.5 g after best supportive care for >= 6 months prior to screening, or Screening 24-hour urinary protein > 3.5 g with at least one high-risk factor defined by the protocol;
4. Estimated glomerular filtration rate (eGFR ) by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formula ≥40 mL/min/1.73 m^2;
5. If taking ACEI(Angiotensin converting enzyme inhibitors), ARB(Angiotensin receptor blocker), a stable dose within 4 weeks before screening is required;
6. Sufficient organ function;
7. Able and willing to provide written informed consent and to comply with the study protocol.

Exclusion Criteria:

1. Participants with a secondary cause of MN;
2. Cyclosporine resistance;
3. Received treatment drugs for membranous nephropathy;
4. Concomitant with other serious diseases；
5. Received live vaccination, major surgery (excluding diagnostic procedures), and participated in other clinical trials within 28 days prior to receiving the first study drug;
6. Patients who are positive for hepatitis B surface antigen (HBsAg) and/or hepatitis B core antibody (HBcAb), with HBV DNA levels above the normal range (HBsAg and/or HBcAb-positive patients require regular HBV DNA testing); patients positive for hepatitis C virus (HCV) antibodies; or patients with a positive human immunodeficiency virus (HIV) serology.
7. Participants with CD4+ T lymphocyte count < 200 cells/μL;
8. Those who have a clear history of tuberculosis or have received anti- tuberculosis treatment;
9. Participants with known history of severe allergic reactions to humanized monoclonal antibodies, MIL62, or Cyclosporine
10. Breastfeeding or pregnant women;
11. Childbearing potential and unwillingness or impossibility to comply with a scientifically acceptable birth-control method
12. Other conditions unsuitable for participation in this study determined by the Investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-06-02 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate at Week 76 | Week 76
  The proportion of participants who achieved complete remission (CR) based on Urine Protein-to-Creatinine Ratio (UPCR) at week 76.

SECONDARY OUTCOMES:
Complete Remission rate at Week 52. | Week 52
  The proportion of participants who achieved CR based on UPCR at week52 (key secondary endpoints)
Overall remission rate at Week 52 and 76. | Week 52 and 76
  The proportion of participants who achieved overall remission(OR) based on UPCR at week 52 and week76.
Complete remission rate and Overall remission rate at Week 24 and 104. | Week 24 and 104
  The proportion of participants who achieved CR and OR based on UPCR at week 24 and week 104.
Complete remission rate and Overall remission rate at Week 24，52，76 and 104. | Week 24，52，76 and 104
  The proportion of participants who achieved CR or OR as assessed by the Investigators based on 24-hour urine protein at week 24, week 52, week 76 and week 104.
Time to Treatment Failure or Relapse after Overall remission | Up to 104 weeks
  Time to Treatment Failure or Relapse after Complete or Partial Remission
Change in efficacy indicators | Baseline to Week 104
  Change in anti-PLA2R Autoantibody Titer, UPCR, eGFR, 24-hour urine protein and ALB
Change in quality of life | Baseline to Week 104
  Mean Change in T-score from Baseline in the EQ5D Scale at Week 104
Percentage of Participants with Adverse Events (AEs) | up to 104 weeks
  Severity Determined According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0
Percentage of Participants with AEs of Special Interest (AESIs) | Up to 104 weeks
Peripheral B-cell Counts at Specified Timepoints | Up to 104 weeks
Serum Concentrations of MIL62 at Specified Timepoints | Up to 104 weeks
Incidence of ADAs during the study | Up to 104 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided